CLINICAL TRIAL: NCT00241826
Title: Prospective Investigation of Pulmonary Embolism Diagnosis III (PIOPED III)
Brief Title: Prospective Investigation of Pulmonary Embolism Diagnosis III
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 329; U01HL077155 (NIH); U01HL077149 (NIH); U01HL077150 (NIH); U01HL077151 (NIH); U01HL077153 (NIH); U01HL077154 (NIH); U01HL077358 (NIH); U01HL081593 (NIH); U01HL081594 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2009-07

CONDITIONS: Lung Diseases; Pulmonary Embolism
MeSH Terms: conditions — Lung Diseases; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Magnetic Resonance Angiography — Participants will undergo magnetic resonance angiography.
Procedure: Magnetic Resonance Venography — Participants will undergo magnetic resonance venography.

SUMMARY:
The purpose of this study is to determine the diagnostic accuracy of gadolinium-enhanced magnetic resonance angiography (Gd-MRA) of the pulmonary arteries in combination with magnetic resonance venography (MRV) of the veins of the thighs in patients with clinically suspected acute pulmonary embolism (PE).

DETAILED DESCRIPTION:
BACKGROUND:

Prospective Investigation of Pulmonary Embolism Diagnosis III (PIOPED III) follows PIOPED I and PIOPED II. PIOPED I was a multicenter trial supported between 1983 and 1989 to evaluate the sensitivity and specificity of two major, widely used technologies, radionuclear imaging (ventilation-perfusion scanning) and pulmonary angiography, for the diagnosis of PE. PIOPED II was a multicenter trial conducted between 2000 and 2005 to determine the value of contrast-enhanced spiral computed tomography (spiral CT) for the diagnosis of acute PE.

In PIOPED II, among 7,284 patients with suspected acute PE, 18.6% had an elevated creatinine, 3.9% were allergic to iodinated contrast material, and 4.7% of women were pregnant. One or more of these relative contraindications to an imaging procedure that would expose the patient to ionizing radiation or iodinated contrast material was present in 24.4% of patients with suspected acute PE. Although patients with relative contraindications often take the risk of CT or digital subtraction angiography (DSA) because of the importance of having a definitive diagnosis, such patients could benefit from safer diagnostic testing with Gd-MRA/MRV if it is shown to be sufficiently accurate.

The purpose of this investigation is to determine the extent to which Gd-MRA/MRV can serve as a diagnostic test in patients with clinically suspected PE and thereby eliminate the need for iodinated contrast material or ionizing radiation in patients who have a relative contraindication to one of them. This is important because 24% of patients with suspected acute PE have a relative contraindication to diagnostic procedures that involve ionizing radiation or iodinated contrast material.

DESIGN NARRATIVE:

PIOPED III is a multicenter prospective investigation designed to determine the diagnostic accuracy of Gd-MRA of the pulmonary arteries in combination with MRV of the veins of the thighs in patients with clinically suspected acute PE. The diagnostic accuracy of Gd-MRA alone and in combination with MRV will be expressed as sensitivity, specificity, and likelihood ratio for positive and negative tests. The study design is a prospective study of consecutive patients incorporating standardized inclusion/exclusion criteria, complete ascertainment of patient characteristics and outcomes, uniform diagnostic criteria, and unbiased paired central readings of imaging studies. Over a period of 2 years, 1,256 patients with suspected acute PE will be recruited at clinical centers. Composite reference standards will be used to diagnose venous thromboembolism (VTE) and exclude PE. It is expected that 314 patients will have acute VTE and they will undergo Gd-MRA/MRV. It is expected that 942 patients will be shown not to have PE. From among this group, 314 patients will be randomly selected for the index test, Gd-MRA/MRV.

ELIGIBILITY:
Inclusion Criteria:

* Acute PE of diagnostic concern
* Informed consent
* Willing to undergo Gd-MRA/MRV

Exclusion Criteria:

* Any implanted ferromagnetic foreign body, including a ferromagnetic cerebral aneurysm clip or implanted electrical device/pump
* Dependency on a continuous connection to an external electrical device/pump (e.g., pacemaker, internal defibrillator, cochlear implant, nerve or bone stimulator implant, ICU appliance) and cardiac pacing wires
* Severe claustrophobia
* Severe shaking
* Inability to lie still for 30 minutes
* Pregnancy and nursing mothers
* Serum creatinine levels within range of normal at local center
* Sickle cell anemia, other hemoglobinopathies, and other hemolytic anemias
* Critical illness, shock or hypotension, hemodynamic instability, ventilatory support, chronic anticoagulation, inferior vena cava filter
* Documented episodes of ventricular fibrillation or sustained ventricular tachycardia within the past 24 hours
* Myocardial infarction within the past month
* History of allergy to gadolinium-containing contrast agents or to iodinated contrast media
* Current symptomatic asthma
* Clinical evidence of venous thrombosis of the upper extremity
* Prisoners
* Institutionalized or mentally handicapped patients
* Too large to fit in MRI unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with suspected acute pulmonary embolism will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1256 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2009-04

PRIMARY OUTCOMES:
Diagnosis or exclusion of pulmonary embolism in agreement with a reference standard | Measured within 36 to 48 hours of study entry

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fowler, PhD, Principal Investigator — George Washington University; Charles Hales, MD, Principal Investigator — Massachusetts General Hospital; Russell Hull, MBBS, MSc, Principal Investigator — University of Calgary; Kenneth Leeper, Jr., MD, Principal Investigator — Emory University; David Naidich, MD, Principal Investigator — NYU Langone Health; Daniel Sak, Do, Principal Investigator — St. Joseph Mercy Oakland; Paul D. Stein, MD, Study Chair — St. Joseph Mercy Oakland; John Weg, MD, Principal Investigator — University of Michigan at Ann Arbor; Pamela Woodard, MD, Principal Investigator — Washington University School of Medicine
Locations (9):
- United States (8):
  - Emory University, Atlanta, Georgia
  - Divison of Lung Diseases, NHLBI, Bethesda, Maryland
  - Data Coordinating Center, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - St. Joseph Mercy-Oakland, Pontiac, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - NYU Medical Center, New York, New York
- Foothills Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Stein PD, Chenevert TL, Fowler SE, Goodman LR, Gottschalk A, Hales CA, Hull RD, Jablonski KA, Leeper KV Jr, Naidich DP, Sak DJ, Sostman HD, Tapson VF, Weg JG, Woodard PK; PIOPED III (Prospective Investigation of Pulmonary Embolism Diagnosis III) Investigators. Gadolinium-enhanced magnetic resonance angiography for pulmonary embolism: a multicenter prospective study (PIOPED III). Ann Intern Med. 2010 Apr 6;152(7):434-43, W142-3. doi: 10.7326/0003-4819-152-7-201004060-00008. PMID 20368649